CLINICAL TRIAL: NCT01735019
Title: Estimating EC95 of Remifentanil for Cough Prevention During Emergence From Total Intravenous Anesthesia With Propofol and Remifentanil in Patients Undergoing Transsphenoidal Hypophysectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2012-0350
Record Dates: First submitted 2012-11-18; First posted 2012-11-28 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2012-11

CONDITIONS: Hypophysectomy
Keywords: EC95, effective concentration in 95% of subjects

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- group 1 (Experimental): administration of remifentanil with target-controlled infusion (TCI) system at a given concentration during anesthetic emergence
  Interventions: Drug: Administration of remifentanil with TCI system

INTERVENTIONS:
Drug: Administration of remifentanil with TCI system — A given effect site concentration of remifentanil would be administered to subjects using TCI system. According to biased coin design, the given concentration of remifentanil is determined according to success or failure of just previously enrolled patient. If the former patient did not cough during anesthetic emergence at a given concentration (success), the next patient will be randomly allocated into the same concentration of remifentanil with 18/19 of probability or the lower concentration of remifentanil by 0.4 ng/ml with 1/19 of probability. If the former patient coughed during anesthetic emergence (failure), the next will be automatically allocated into the higher concentration of remifentanil by 0.4 ng/ml.

SUMMARY:
In patients undergoing hypophysectomy through transsphenoidal approach, preventing cough during anesthetic emergence is important to avoid hemorrhage and cerebrospinal fluid leakage. Previous reports demonstrated that administration of remifentanil during anesthetic emergence could reduce the incidence and severity of cough during anesthetic emergence. Therefore, the objective of this study is to determine EC95 of remifentanil for preventing cough during anesthetic emergence in patients undergoing hypophysectomy with transsphenoidal approach.

ELIGIBILITY:
Inclusion Criteria:

* scheduled to undergo hypophysectomy with transsphenoidal approach
* American Society of Anesthesiologists physical status I or II
* more than 20 years old

Exclusion Criteria:

* acute or chronic respiratory disease
* uncontrolled hypertension
* taking sedatives or anti-tussive
* gastro-esophageal reflux
* pregnant or breast feeding
* patients who cannot understand statements for subjects or this study itself

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The occurrence of cough during anesthetic emergence | 5 min after extubation
  At a given effect-site concentration of remifentanil, if cough does not occur during anesthetic emergence, it would be considered as a success. On the other hand, if cough occurs during anesthetic emergence, it would be considered as a failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea